CLINICAL TRIAL: NCT01063920
Title: A Double-Blind, Double-Dummy, Randomized, Active-Comparator, Non-Inferiority Study of LT-NS001 Versus Naprosyn® for Twelve Weeks in Osteoarthritis Patients to Compare Endoscopic Gastric Ulcer Rates
Brief Title: Rates of Gastric Ulcer by Endoscopy in Knee Osteoarthritis Patients Receiving LT-NS001 Versus Naprosyn®
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Logical Therapeutics (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: K. Lea Sewell, M.D./Vice President Clinical Development, Logical Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LT-NS001-003
Record Dates: First submitted 2010-01-29; First posted 2010-02-05 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Osteoarthritis
Keywords: LT-NS001; Gastric Ulcers; NSAID; Osteoarthritis; Naproxen
MeSH Terms: conditions — Osteoarthritis; Stomach Ulcer | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- LT-NS001 (Experimental): LT-NS001 1200 mg b.i.d. p.o. for 12 weeks
  Interventions: Drug: LT-NS001
- Naprosyn® (Active Comparator): Naprosyn® 500 mg b.i.d for 12 weeks
  Interventions: Drug: Naprosyn®

INTERVENTIONS:
Drug: LT-NS001 — 1200 mg b.i.d. p.o. for 12 weeks
  Arms: LT-NS001
Drug: Naprosyn® — 500 mg b.i.d. p.o. for 12 weeks
  Arms: Naprosyn®

SUMMARY:
LT-NS001 is a prodrug of Naproxen, which is inactive as a cox inhibitor while intact and is rapidly metabolized to Naproxen once absorbed. This trial will compare the rate of gastric ulcer by endoscopy over three months in patients with knee osteoarthritis, with patients receiving either LT-NS001 at a dose which provides comparable dose levels of Naproxen, or Naprosyn® 500mg (an approved treatment for OA).

DETAILED DESCRIPTION:
This is a double-blind, double-dummy, active-comparator study of LT-NS001 versus Naprosyn® for 12 weeks in patients aged 45-80 with osteoarthritis of the knee who are candidates for ongoing NSAID therapy. The percentage of patients with a gastric ulcer by endoscopy (EGD) at week 12 will be compared. EGD is performed at screening and months 1, 2, and 3. Secondary objectives include assessment of pain in the affected knee by WOMAC questionnaire to demonstrate non-inferior pain control using LT-NS001 as compared to Naprosyn®. Information about gastrointestinal pain and tolerability will be collected.

The length of the study is up to 19 weeks with a 2-3 week screening period, a 12 week treatment period and a 4 week post treatment monitoring period.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of knee
* Appropriate candidate for chronic NSAID therapy due to moderate or severe pain on most days in the 28 days before screening for study.

Exclusion Criteria:

* Pregnant/Nursing women
* History of GI bleeding, perforation or obstruction
* A documented symptomatic GI ulcer during past 5 years
* Presence of GI ulcer or more than 2 erosions on screening endoscopy
* Allergy to naproxen (or naproxen intolerance), acetylsalicylic acid, or other NSAID drug

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Gastric Ulcer by Endoscopy | Baseline, Day 29, Day 57 and Day 85

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Screening, Baseline, Days 15, 29, 57 and 85
Population pharmacokinetic analysis will assess the influence of covariates on the absorption/metabolism of LT-NS001 to naproxen | Two separate days after Day 14, at least two weeks apart

CONTACTS AND LOCATIONS:
Overall Officials: Jay L Goldstein, MD, Principal Investigator — University of Illinois at Chicago, Department of Medicine
Locations (65):
- United States (65):
  - Greystone Medical Research, LLC, Birmingham, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Radiant Research, Chandler, Arizona
  - Dedicated Clinical Research Inc., Surprise, Arizona
  - Radiant Research Inc., Tucson, Arizona
  - Adobe Gastroenterology Research, LLC, Tucson, Arizona
  - Genova Clinical Research Inc., Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Orange County Clinical Trials, Anaheim, California
  - Theresa Sligh, MD, Burbank, California
  - Torrance Clinical Research, Lomeita, California
  - West Gastroenterology Associates, Los Angeles, California
  - Facey Medical Center, Mission Hills, California
  - Desert Medical Group, Palm Springs, California
  - Medical Affiliated Research Center Inc., San Diego, California
  - Cynthia Schaeffer, MD, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Eastern Clinical Research Unit, Hialeah, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Drug Study Institute, Jupiter, Florida
  - University Clinical Research Inc., Pembroke Pines, Florida
  - Radiant Research, Pinellas Park, Florida
  - Accord Clinical Research LLC, Port Orange, Florida
  - Miami Research Associates, South Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Gold Coast Research LLC, Weston, Florida
  - Thomas Schnitzer, MD, Chicago, Illinois
  - Welborn Clinic, Evansville, Indiana
  - MediSphere Medical Research Center LLC, Evansville, Indiana
  - Venture Resource Group Inc., Mission, Kansas
  - Pinnacle Medical Research, Overland Park, Kansas
  - Delta Research Partners LLC, Bastrop, Louisiana
  - SNBL Clinical Pharmacology Center, Baltimore, Maryland
  - Metropolitan Gastroenterolgy Group PC, Chevy Chase, Maryland
  - Arthritis and Osteoporosis Cener of Maryland, Frederick, Maryland
  - MidAtlantic Medical Research Centers/Bean Medical Center, Hollywood, Maryland
  - Dynamic Clinical Research, Kansas City, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Montana Health Research Institute Inc., Billings, Montana
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Affiliated Clinical Research Inc., Las Vegas, Nevada
  - Clifton-Wallington Medical Group, Clifton, New Jersey
  - Research Across America, New York, New York
  - Allergy Asthma Immunology of Rochester Research Center, Rochester, New York
  - Carolina Digestive Health Associates PA, Charlotte, North Carolina
  - Peters Medical Research LLC, High Point, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Radiant Research-Akron, Akron, Ohio
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Clinical Research Associates LLC, Oklahoma City, Oklahoma
  - Keith Klatt, MD, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Corsicana Medical Research PLLC, Corsicana, Texas
  - Galenos Research, Dallas, Texas
  - Clinical Trial Network, Houston, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - Quality Research Inc., San Antonio, Texas
  - Arthritis and Osteoporosis Clinic Research Center of Central Texas, Waco, Texas
  - Physicians Research Options LLC, Draper, Utah